CLINICAL TRIAL: NCT06405945
Title: Evalutaion of the SNPs Test in Average Cervical Cancer Screening Episode
Brief Title: Cervical Cancer Susceptible Population Classification
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Wila-Cer-01
Record Dates: First submitted 2024-05-05; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cervical Cancer Susceptible Population Classification
MeSH Terms: interventions — Polymerase Chain Reaction; Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal: HPV negative， TCT negative
  Interventions: Genetic: PCR and sequence
- LSIL: HPV postive, TCT: CIN I or Colposcopy LSIL
  Interventions: Genetic: PCR and sequence
- HSIL: HPV postive, TCT: CIN II-III or Colposcopy HSIL
  Interventions: Genetic: PCR and sequence
- cervical cancer: HPV positive, Histopathology: cervical cancer
  Interventions: Genetic: PCR and sequence

INTERVENTIONS:
Genetic: PCR and sequence — sequence the mutatation SNPs

SUMMARY:
Cervical cancer is the third most common lethal tumor globally, causing around a quarter million deaths annually, despite the availability of HPV vaccines. Recent Genome-wide association studies (GWAS) have identified numerous genetic markers linked to cervical cancer, including rs10175462, rs10007915, rs35721900, and rs61646675, which have been verified as being related to susceptibility to cervical cancer. However, many reports lack clarity, consistency, and validation. In this comprehensive study, we will analyze the genomic risk factors associated with cervical cancer, classify individuals into different risk categories, and explore potential biomarkers and therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged >=18 years at time of consent
2. Intended to undergo screening colposcopy
3. Considered by a physician or healthcare provider as being of "average risk" for cervical cancer
4. Willing to consent to blood draw cervical disease treatments
5. Willing to sonsent to follow-up for five years as per protocol

Exclusion Criteria:

1. History of cervical cancer
2. History of any malignancy (patients who have undergone surgical removal of skin squamous cell cancer may be enrolled provided the procedure was completed at least 12 months prior to the date of provision of informed consent for the study)
3. Currently taking any anti-neoplastic or disease-modifying anti-rheumatic drugs.
4. Any major physical trauma (e.g. disruption of tissue, surgery, organ transplant, blood product transfusion) within the 30 days leading up to the provision of informed consent
5. Known medical condition which, in the opinion of the investigator, should preclude enrollment into the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HPV positive person at average risk of cervical cancer
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2034-04-30 (Estimated); Study Completion 2036-06 (Estimated)

PRIMARY OUTCOMES:
Evalutaiton of the SNPs test in an average cervical cancer patients screening episode | two years

SECONDARY OUTCOMES:
Classified susceptied person into different ladders | two years

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Wang, Doctor, Study Chair — The First Affiliated Hospital of USTC
Locations (1):
- The First Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided